CLINICAL TRIAL: NCT03527511
Title: Effect of Active Vitamin D and Etelcalcetide on Human Osteoclasts in Patients With Chronic Kidney Disease
Acronym: RENOCLASTE
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL17_0785; 2017-A03241-52 (Other: ID-RCB)
Record Dates: First submitted 2018-04-19; First posted 2018-05-17 (Actual); Last update posted 2020-03-31 (Actual); Status verified 2020-03

CONDITIONS: Bone Disorder; Chronic Kidney Diseases
MeSH Terms: conditions — Bone Diseases; Renal Insufficiency, Chronic

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Samples specific to the study (urea, creatininemia, CA²+, Phosphorus, PTH, Alkaline phosphatase, vitamin D) will be collected and analyzed as part of the usual care. An additional 20 mL blood is collected for analysis of osteoclastogenesis
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Measure of etecalcetide on osteoclastic biology — In vitro evaluation of osteoclastic biology after blood sampling of patients.

SUMMARY:
The optimal management of mineral and bone disorders associated to chronic kidney disease (CKD-MBD) is a daily challenge for nephrologists. Its consequences may be immediate (biological abnormalities such as hypocalcemia, hyperphosphatemia, hyperparathyroidism, etc.) or delayed (fractures, renal osteodystrophy, vascular calcifications, increased morbi-mortality and growth retardation in the youngest patients). CKD-MBD is defined by the association of one or more of the following abnormalities: 1/ disturbances in calcium, phosphate, PTH or vitamin D metabolism, 2/ bone and growth abnormalities, and 3/ calcifications of vessels or soft tissues .

Three main bone characteristics can be modified by CKD, namely turnover, mineralization and volume. They should therefore be carefully assessed to distinguish between the different sub-types of renal osteodystrophy, as defined in the 2006 K-DIGO guidelines on the TMV classification . The primary bone lesion in pediatric CKD, at least in pediatric patients reaching end-stage renal disease without any previous management, is the high-turnover/hyperparathyroidism, because of high circulating PTH levels with low 1-25 vitamin D levels. Conversely, low turnover (or adynamic bone) may be observed in dialysis children receiving too much calcium and/or vitamin D analogs. All these lesions are deleterious on the long-term, increasing both the risk of growth retardation, fractures and vascular calcifications .

In order to better understand the complex pathophysiology of renal osteodystrophy, biomarkers of bone and phosphate/calcium metabolism may be used, but their interpretation may be challenging in the context of CKD. The gold standard remains bone biopsy at the iliac crest with histomorphometry, but it is rarely performed in Europe .

The research team of this study has developed and validated a unique non-invasive technique to differentiate circulating human monocytes into mature and functional osteoclasts, using only 15 mL of total blood (instead of conventional techniques they used to use, with 200 to 250 mL of total blood). They propose to use this innovative tool in the specific setting of CKD.

The current management of CKD-MBD consists mainly of correcting native vitamin D deficiency, decreasing phosphate levels (using nutritional management and phosphate-binders), and decreasing PTH levels (using active vitamin D, calcimimetics such as cinacalcet and etelcalcetide, and/or surgical parathyroidectomy) . Active vitamin D analogs and calcimimetics are cornerstone of this management.

The first working hypothesis is the following: when CKD progresses and glomerular filtration rate (GFR) decreases, 1-25-D is able to inhibit osteoclastic differentiation, however to a lesser extent to what is observed in healthy controls with normal renal function.

The second working hypothesis is therefore the following: etecalcetide could be an inhibitor of osteoclastic resorption and a stimulator of osteoblastogenesis. When CKD worsens and GFR decreases, etelcalcetide inhibits osteoclastic differentiation, however to a lesser extent to what is observed in subjects with normal renal function.

Aims In Vitro

1. Effects of 1-25-D and etecalcetide on human osteoclastogenesis and osteoclastic resorption (in cells obtained from CKD patients at different stages of CKD)
2. Effects of 1-25-D and etecalcetide on murine osteoblastogenesis and mineralization

ELIGIBILITY:
Inclusion Criteria:

* Child of age> 2 years old and <18 years old.
* Child over 10 kg having a blood sample as part of the treatment (due to regulatory constraints for blood volume taken by 30-day period of 40 mL in children over 10 kg)
* Child with chronic kidney disease followed in the pediatric nephrology department of the "Hôpital Mère Enfant" in Bron.
* Child and parent / holder of parental authority who has been informed of the study and does not object to participate

Exclusion Criteria:

* Bone damage associated with genetic renal disease known to induce specific bone involvement: oxalosis, cystinosis, Pierson syndrome, paracellin mutation, dominant polycystic disease
* Treatment in progress that may have a specific impact on the bone: growth hormone, bisphosphonates, teriparatide.

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: 35 children with chronic kidney disease (CKD). 5 children per CKD group: CKD stage 1, stage 2, stage 3, stage 4, stage 5, dialysis, transplantation.
Sampling Method: Non-Probability Sample
Enrollment: 21 (Actual)
Dates: Start 2018-05-14 (Actual); Primary Completion 2018-10-22 (Actual); Study Completion 2018-10-22 (Actual)

PRIMARY OUTCOMES:
Active vitamin D action on osteoclasts | 1 day
  Patients' cells will be used to ex vivo. Osteoclastic biology will be analyzed according to two components: differentiation and resorption activity.
Etecalcetide action on osteoclasts | 1 day
  Patients' cells will be used to ex vivo. Osteoclastic biology will be analyzed according to two components: differentiation and resorption activity.

CONTACTS AND LOCATIONS:
Locations (1):
- Service de Néphrologie, Rhumatologie et Dermatologie Pédiatriques - Hôpital Femme Mère Enfant - Bron., Bron, France

IPD SHARING:
Plan to Share IPD: No